CLINICAL TRIAL: NCT01102075
Title: The Effect of Low Frequency Electroacupuncture on Waist Circumference in Obesity-Three Arm Randomized Controlled Trial, Pilot Study
Brief Title: The Effect of Electroacupuncture on Obesity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Sung Keel Kang, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KOMC MIRB 2009-6
Record Dates: First submitted 2010-04-06; First posted 2010-04-12 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2009-09

CONDITIONS: Obesity
Keywords: Obesity; Electroacupuncture; Sham electroacupuncture; Waist circumference; Thickness of subcutaneous fat
MeSH Terms: conditions — Obesity | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Electroacupuncture (Experimental): The Electroacupuncture therapy protocol included a total of 12 acupuncture points at the CV12,CV6, bilateral ST25, SP15, SP14,LI4, LI11, ST36, ST44. All acupuncture points were prepared with 70% alcohol pads, and disposable stainless steel needles were used. Abdominal acupuncture points were inserted horizontally 6~6.5cm in depth and the others were inserted vertically 2~2.5cm in depth until patient can feel De-Qi. All acupuncture points were stimulated electrically with a frequency of 24 Hz an intensity of 0.27-1.3mA(tolerable strength) with continuous stimulation by the pulse generator. The participants were given treatment twice a week for 30 minutes for 5 weeks by practitioner who had had 6 years of acupuncture training and 3 more years of clinical experience.
  Interventions: Device: Electroacupuncture
- Sham electroacupuncture procedure (Sham Comparator): The Sham electroacupuncture therapy protocol(Non-acupoint, No electrical stimulation)included the same number and type of needle, duration, frequency of sessions and practitioner as for the EA treatment, but superficially at non acupuncture points 15 mm to the lateral of each acupuncture point was treated. The points were not stimulated electrically, but the sound of the pulse generator was heard by the participants. (Lee SH, LeeBC 2009) Those receiving EA or SEA therapy were treated on alternate days to prevent crosstalk among groups, which could have compromised the blinded study design.
  Interventions: Device: Sham electroacupuncture procedure
- Waiting list (No Intervention): No treatment was done for waiting group, but could receive same treatments as Electroacupuncture group after the end of trial.

INTERVENTIONS:
Device: Electroacupuncture — We used Electrical stimulator(STN-111,Stratek)with a frequency of 24 Hz and intensity of 0.27-1.3mA(tolerable strength), asymmetric interactive pulse with continuous stimulation by the pulse generator. The participants were given treatment twice a week for 30 minutes for 5 weeks(10 sessions) by practitioner.(n=13)
  Other Names: EA group
  Arms: Electroacupuncture
Device: Sham electroacupuncture procedure — We used same electroacupuncture device, number and type of needle, duration, frequency of sessions and practitioner as for the EA treatment. Specific details are as described in the arm description.(n=13)
  Other Names: Sham EA group
  Arms: Sham electroacupuncture procedure

SUMMARY:
The purpose of this study is to determine whether electroacupuncture is effective on waist circumference in obesity.

DETAILED DESCRIPTION:
Many studies have reported on the beneficial effects of acupuncture for obesity, although some negative reports also existed.(Wang F. et al. 2008)Recently conducted systematic review of Pittler and Ernst reported that there was insufficient, but not conclusive evidence to support the efficacy of acupuncture and acupressure for weight loss. However, most of these studies had methodological limitation, such as lack of adequate control group or unclear specific effect of electroacupuncture alone because auricular acupuncture was administered as well. In this sudy, we had three-arm randomized controlled trial(with sham control group) to investigate whether electroacupuncture is effective in the treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference: Male>= 90 cm, Female >= 85 cm
* BMI over than 25kg/m2

Exclusion Criteria:

* Secondary obesity caused by endocrine disease, e.g., polycystic ovary syndrome, diabetes mellitus, Cushing's syndrome, hypothyroidism etc.
* Heart disease,e.g.,arrhythmia, heart failure, myocardial infarction, and patient with pacemaker
* Hypertension, hyperlipidemia or hypercholesterinemia patients on medication
* Stroke or otherwise unable to exercise
* Pregnant or lactating women
* Childbirth within 6 months
* Management for weight control within 3 months
* Any other conditions deemed unsuitable for trial as evaluated by the physician-in-charge

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
waist circumference | At 5 weeks (post treatment)

SECONDARY OUTCOMES:
Thickness of abdominal subcutaneous fat | Study Day 1 (Baseline)
  Thickness of abdominal subcutaneous fat was measured by digital skinfold caliper(FatTrack).
Thickness of abdominal subcutaneous fat | At 3weeks
  Thickness of abdominal subcutaneous fat was measured by digital skinfold caliper(FatTrack).
Thickness of abdominal subcutaneous fat | At 5weeks (post treatment)
  Thickness of abdominal subcutaneous fat was measured by digital skinfold caliper(FatTrack).
Thickness of abdominal subcutaneous fat | At 8weeks after first treatment (follow up)
  Thickness of abdominal subcutaneous fat was measured by digital skinfold caliper(FatTrack).
Waist hip ratio | Study Day 1 (Baseline)
Waist hip ratio | At 3weeks
Waist hip ratio | At 5weeks (post treatment)
Waist hip ratio | At 8weeks after first treatment (follow up)
Body Mass Index | Study Day 1 (Baseline)
  Body Mass Index was measured by Inbody 720
Body Mass Index | At 3weeks
  Body Mass Index was measured by Inbody 720
Body Mass Index | At 5weeks (post treatment)
  Body Mass Index was measured by Inbody 720
Body Mass Index | At 8weeks after first treatment (follow up)
  Body Mass Index was measured by Inbody 720
Body fat ratio | Study Day 1 (Baseline)
  Body fat ratio was measured by Inbody 720
Body fat ratio | At 3weeks
  Body fat ratio was measured by Inbody 720
Body fat ratio | At 5weeks (post treatment)
  Body fat ratio was measured by Inbody 720
Body fat ratio | At 8weeks after first treatment (follow up)
  Body fat ratio was measured by Inbody 720
Visceral Fat Area | Study Day 1 (Baseline)
  Visceral Fat Area was measured by Inbody 720
Visceral Fat Area | At 3weeks
  Visceral Fat Area was measured by Inbody 720
Visceral Fat Area | At 5weeks (post treatment)
  Visceral Fat Area was measured by Inbody 720
Visceral Fat Area | At 8weeks after first treatment (follow up)
  Visceral Fat Area was measured by Inbody 720
Body weight | Study Day 1 (Baseline)
  Body weight was measured by Inbody 720
Body weight | At 3weeks
  Body weight was measured by Inbody 720
Body weight | At 5weeks (post treatment)
  Body weight was measured by Inbody 720
Body weight | At 8weeks after first treatment (follow up)
  Body weight was measured by Inbody 720
Obesity degree | Study Day 1 (Baseline)
  Obesity degree was measured by Inbody 720
Obesity degree | At 3weeks
  Obesity degree was measured by Inbody 720
Obesity degree | At 5weeks (post treatment)
  Obesity degree was measured by Inbody 720
Obesity degree | At 8weeks after first treatment (follow up)
  Obesity degree was measured by Inbody 720
Bulimia Test Revised | Study Day 1 (Baseline)
Bulimia Test Revised | At 5weeks (post treatment)
Korean version of Obesity-related QOL scale | Study Day 1 (Baseline)
Korean version of Obesity-related QOL scale | At 5weeks (post treatment)
Body Shape Questionnaire | Study Day 1 (Baseline)
Body Shape Questionnaire | At 5weeks (post treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Keel Kang, Doctor, Principal Investigator — Kyunghee University Medical Center Oriental Hospital
Locations (1):
- Kyunghee University Medical Center, Seoul, Hoegi-dong, Dongdaemun-gu, South Korea

REFERENCES:
- [Background] Lee SH, Lee BC. Electroacupuncture relieves pain in men with chronic prostatitis/chronic pelvic pain syndrome: three-arm randomized trial. Urology. 2009 May;73(5):1036-41. doi: 10.1016/j.urology.2008.10.047. PMID 19394499
- [Background] Wang F, Tian DR, Han JS. Electroacupuncture in the treatment of obesity. Neurochem Res. 2008 Oct;33(10):2023-7. doi: 10.1007/s11064-008-9822-6. Epub 2008 Aug 22. PMID 18719995
- [Background] Pittler MH, Ernst E. Complementary therapies for reducing body weight: a systematic review. Int J Obes (Lond). 2005 Sep;29(9):1030-8. doi: 10.1038/sj.ijo.0803008. PMID 15925954